CLINICAL TRIAL: NCT01549457
Title: The Effect of Weekly Text-message Communication on Treatment Completion Among Patients With Latent Tuberculosis Infection: a Randomised Controlled Trial (WelTel LTBI)
Brief Title: TB mHealth Study - Use of Cell Phones to Improve Compliance in Patients on LTBI Treatment
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H11-02216
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Latent Tuberculosis Infection
Keywords: latent tuberculosis; text message interventions; medication adherence
MeSH Terms: conditions — Latent Tuberculosis; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-intervention (No Intervention): Participants will only receive standard of care
- Cell phone intervention arm (Experimental): Upon consent, participants will be randomly assigned to receive either 1) standard of care (9 months of INH or 4 months of RIF) and weekly SMS text messages via mobile phone or 2) standard of care (9 months of INH or months of RIF) without weekly SMS text messages via mobile phone.
  Interventions: Other: Cell phone text messages

INTERVENTIONS:
Other: Cell phone text messages — Participants in the intervention arm will receive weekly text messages from the TB control clinic asking how they are.
  Arms: Cell phone intervention arm

SUMMARY:
This study will examine the impact of use of mobile phones and text messaging on adherence to treatment for patients with latent TB infection. Half (50%) of the 350 anticipated study participants will receive weekly text messages inquiring on their health status in relation to their prescribed treatment, while the other half (50%) will not receive weekly text messages at all. Medical adherence will be assessed by monthly blood-work, clinic visits and by interviewing patients at each of these visits.

The investigators hypothesis is that enhanced communication with a health care provider, via a structured cell phone SMS text messaging based program (WelTel), will result in a 15% improvement in the proportion of patients who successfully complete their LTBI treatment regimens.

DETAILED DESCRIPTION:
1. Purpose

   The purpose of this study is to compare the proportion of patients who are adherent to their TB medications among those receiving weekly text messages plus standard of care and those who receive standard of care only.
2. Justification:

   Previous research has shown that weekly text messages from a health care provider increases medication adherence for HIV patients. The investigators would like to determine if a similar effect in terms of adherence can be seen in patients receiving medication for latent tuberculosis infection
3. Objectives

Primary Objective:

1) To compare successful treatment completion rates for patients treated with 9 months of INH or 4 months of RIF between those receiving weekly SMS text messages via mobile phone plus standard of care to those receiving standard care. The standard of care at the TB clinics for all LTBI patients includes provision of a 30 day supply of medications - isoniazid 300mg daily for 9 months months or rifampin 600mg daily for 4 months - at a time, monthly blood-work and monthly clinic visits. Successful treatment completion is defined as taking at least 80% of the doses of INH prescribed within 12 months or at least 80% of the doses of RIF prescribed within 6 months.

Secondary Objectives:

1. To compare the proportion of prescribed doses taken on schedule (daily adherence) prior to medication discontinuation or interruption on medical advice between those receiving weekly SMS text messages via mobile phone to those receiving standard care;
2. To measure patient satisfaction with the SMS intervention using a provider administered questionnaire including a series of Likert questions.

4) Research Method

This study is a prospective open-label multicentre randomized controlled trial of a clinical intervention. It is estimated that 350 study participants will be required to have 80% power to detect a 15% difference in adherence at a .05 level of significance. In addition to recruiting English-speaking participants, the investigators will also be recruiting participants that have Chinese and Punjabi as their first language.

Upon consent, participants will be randomly assigned to receive either 1) standard of care (9 months of INH or 4 months of RIF) and weekly SMS text messages via mobile phone or 2) standard of care (9 months of INH or 4 months of RIF) without weekly SMS text messages via mobile phone.

The clinicians, pharmacists and researchers involved in evaluating compliance will not be blinded to the allocation of the intervention and control groups, as they will be required to review patients charts periodically, respond to patients text messages when they are experiencing difficulty in taking medications or side effects, as well as to ensure the successful operation of the SMS technology platform.

ELIGIBILITY:
Inclusion Criteria:

1. Are initiating treatment for latent TB infection;
2. Are over the age of 18 years old;
3. Own a mobile phone or share access mobile phone access with a household member who consents to participate; AND
4. Demonstrate sufficient ability to communicate via text messaging in English or have a family member or friend that is able to provide translation and assistance with text messaging for the duration of the study

Exclusion Criteria:

1. Individuals under the age of 18;
2. Unable to adequately send and receive text messages for any reason OR
3. Enrolled in another clinical trial that may assess or influence treatment adherence.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Successful completion of LTBI treatment regimens. | 4 or 9 months
  Successful treatment completion is defined as taking at least 80% of the doses of INH prescribed within 12 months or at least 80% of RIF prescribed within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Richard Lester, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - New Westminster TB Control Clinic, New Westminster, British Columbia
  - Vancouver Downtown TB Control Clinic, Vancouver, British Columbia
  - Vancouver TB Control Clinic (VTC),, Vancouver, British Columbia

REFERENCES:
- [Derived] El Joueidi S, Bardosh K, Musoke R, Tilahun B, Abo Moslim M, Gourlay K, MacMullin A, Cook VJ, Murray M, Mbaraga G, Nsanzimana S, Lester R. Evaluation of the implementation process of the mobile health platform 'WelTel' in six sites in East Africa and Canada using the modified consolidated framework for implementation research (mCFIR). BMC Med Inform Decis Mak. 2021 Oct 26;21(1):293. doi: 10.1186/s12911-021-01644-1. PMID 34702229
- [Derived] Johnston JC, van der Kop ML, Smillie K, Ogilvie G, Marra F, Sadatsafavi M, Romanowski K, Budd MA, Hajek J, Cook V, Lester RT. The effect of text messaging on latent tuberculosis treatment adherence: a randomised controlled trial. Eur Respir J. 2018 Feb 7;51(2):1701488. doi: 10.1183/13993003.01488-2017. Print 2018 Feb. PMID 29437940
- [Derived] van der Kop ML, Memetovic J, Patel A, Marra F, Sadatsafavi M, Hajek J, Smillie K, Thabane L, Taylor D, Johnston J, Lester RT. The effect of weekly text-message communication on treatment completion among patients with latent tuberculosis infection: study protocol for a randomised controlled trial (WelTel LTBI). BMJ Open. 2014 Apr 9;4(4):e004362. doi: 10.1136/bmjopen-2013-004362. PMID 24719431